CLINICAL TRIAL: NCT01863121
Title: A Prospective Validation of Child-Turcotte-Pugh-Kumar (CTPK) Score in Predicting Short Term Mortality in Patients With Liver Cirrhosis
Brief Title: Validation of Child-Turcotte-Pugh-Kumar (CTPK) Score in Predicting Short Term Mortality in Patients With Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ashish Kumar, Associate professor & Consultant, Sir Ganga Ram Hospital
Other Study IDs: EC/04/13/503
Record Dates: First submitted 2013-05-21; First posted 2013-05-27 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Cirrhosis
Keywords: cirrhosis; CTPK; CTP; MELD; Severity Score
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cirrhotic Patients: Patients of cirrhosis

SUMMARY:
The CTP score is one of the best proved severity score in predicting mortality in patients with cirrhosis. Portal hypertension and variceal bleed are significant causes of morbidity and mortality in patients with cirrhosis. The recently published CTPK score included variceal variceal bleed status to the CTP score which improved the accuracy of CTP score in predicting short term mortality. CTPK score needs prospective validation.

DETAILED DESCRIPTION:
Once patients with cirrhosis experience decompensation, early mortality risk increases sharply. Child-Pugh score has been the reference for many years for assessing the prognosis of cirrhosis. The model for end-stage liver disease (MELD) score, which was originally designed for assessing the prognosis of cirrhotic patients undergoing transjugular intrahepatic portosystemic shunt (TIPS), is a continuous score relying on three objective variables. Both CTP and MELD scores do not have portal hypertension as one of the parameters. The investigators already know that portal hypertension is also an independent prediction of mortality in patients of cirrhosis, however, both these scores fail to include portal hypertension component in prediction of mortality.

A new severity score was devised by us by modifying existing CTP Score adding to it the endoscopy parameter. The investigators modified the CTP score by adding the points for variceal bleed status of the patients as follows: history of variceal bleed present - 3 points; no history of variceal bleed but large (grade III-IV) varices present - 2 points; and no history of variceal bleed with small (grade I-II) or absent varices - 1 point. These points were added to the conventional CTP score to obtain the CTPK score (maximum score 18, minimum 6). CTPK score is a simple clinical tool and can be calculated at the bedside. It includes the component of portal hypertension, which is not present in the CTP score.

In a retrospective study conducted by the Principal Investigator the CTPK score was found to better predict the short term mortality (1 week, 2 week mortality regardless of treatment) in patients of cirrhosis. It performs significantly better than the CTP score in predicting early mortality, especially at 1 and 2 weeks in cirrhotics. Further prospective validation of this score was warranted. Hence this study aims to prospectively validate the CTPK score for predicting short term mortality in a cohort study of cirrhosis admitted in Sir Ganga Ram Hospital.

STUDY OBJECTIVE

Comparison of CTP score, MELD score with new CTPK score in predicting the mortality at 1 week (primary objective), and at 2 weeks, 1 month, 2 months, 3 months and 6 months (secondary objectives), regardless of the treatment offered.

Primary objective Prediction of short term mortality (1 week)

Secondary objective Prediction of long term mortality 2 weeks, 1 month, 2 months, 3 months and 6 months

All patients of cirrhosis of liver who are admitted in department of gastroenterology & hepatology (Unit - 1, either as inpatient or day care), Sir Ganga Ram Hospital for any reason will be enrolled in study after taking consent & who fit in inclusion criterion. The patients will be subjected to routine evaluation for etiology of cirrhosis and its complications. Severity assessment of cirrhosis will be done by CTP score, MELD score and in addition by new CTPK score. Patients will be treated as per discretion of treating physician. Then patients will be followed up for 6 months at defined intervals. The follow up will be taken as per following time intervals: 1 week, 2 week, 1 month, 2 months 3 months and 6 months. The only parameter assessed in follow up will be their survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient of cirrhosis
* Age between 18 - 75 years
* Admitted in Unit 1 Department of Gastroenterology & Hepatology
* Patients/ LAR who are willing to give written informed consent

Exclusion Criteria:

* Patients with significant cardiopulmonary illness
* Any malignancy including HCC (Hepatocellular Carcinoma)
* Patients who refuse to give consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient of cirrhosis Age between 18 - 75 years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
1-week Survival | 1 week
  Severity assessment of cirrhosis will be done by CTP score, MELD score and in addition by CTPK score. Patients will be treated as per discretion of treating physician. Survival will be assessed at 1 week

SECONDARY OUTCOMES:
2-week Survival | 2 weeks
1-month Survival | 1 month
2-month Survival | 2 months
3-month Survival | 3 months
6-month Survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashish kumar, M..D, Principal Investigator — Department of Gastroenterology & Hepatology, Sir Ganga Ram Hospital; Anil Arora, M.D, Principal Investigator — Department of Gatroenterology & Hepatology, Sir Gnaga Ram Hospital; Praveen Sharma, M.D, Principal Investigator — Department of Gastroenterology & Hepatology, Sir Ganga Ram Hospital; Pankaj tyagi, M.D, Principal Investigator — Department of Gastroenterology & Hepatology, Sir Ganga Ram Hospital
Locations (1):
- Department of Gastroenterology & Hepatology, Sir Ganga Ram Hospital, New Delhi, India

REFERENCES:
- [Background] Kumar A, Sharma P, Sarin SK. Adding variceal status to Child-Turcotte-Pugh score improves its performance in predicting early mortality in cirrhosis: the Child-Turcotte-Pugh-Kumar score. Eur J Gastroenterol Hepatol. 2012 Nov;24(11):1348-9. doi: 10.1097/MEG.0b013e3283579475. No abstract available. PMID 23022921